CLINICAL TRIAL: NCT04745728
Title: Different Immunosuppressive Treatment in Idiopathic Membranous Nephropathy: a Prospective Cohort
Brief Title: Different Immunosuppressive Treatment in iMN
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: iMN cohort
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Idiopathic Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Prednisone; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyclophosphamide and prednisone (Active Comparator): Prednisone will be given at 1mg/kg/d p.o. and will be tapered after 2 months and discontinued over a 6-12 month period.
  Cyclophosphamide will be given at 1-2mg/kg/d p.o. with a target accumulated dose of 12g.
  Azathioprine or mycophenolate mofetil are optional which could be given for a short period of time (<6 months）after discontinuation of cyclophosphamide if patients do not remit at 6 month.
  Interventions: Drug: Prednisone; Drug: Cyclophosphamide
- Rituximab (Active Comparator): Rituximab 1000mg I.V. on Day1 and at 6 month. After 6 months, in patients with response but without complete remission, Rituximab could be stopped or repeated with a 6 month-interval (12 month, 18 month, 24 month) until complete remission. Rituximab 1000mg I.V. will be given on the 15th day after each Rituximab infusion if CD19+ B cell count>5/ul on the 15th day.
  Calcineurin inhibitors (CNI) are optional but should be tapered after 6 months and discontinued after 9 months.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Prednisone — 1mg/kg/d p.o.which will be tapered after 2 months and discontinued over a 6-12 month period.
  Arms: cyclophosphamide and prednisone
Drug: Cyclophosphamide — 1-2mg/kg/d p.o. with a target accumulated dose of 12g.
  Other Names: CTX
  Arms: cyclophosphamide and prednisone
Drug: Rituximab — 1000mg I.V. on D1 and at 6 month. After 6 month, in patients with response but not complete remission, Rituximab could be stopped or repeated with a 6 month-interval (12 month, 18 month, 24 month) until complete remission. Rituximab 1000mg I.V. will be repeated on the 15th day of each Rituximab infusion if CD19+ B cell count>5/ul.
  Other Names: CD20 antibody
  Arms: Rituximab

SUMMARY:
The primary objective of this study is to compare the 24 month remission of different immunosuppressive therapies in the treatment of idiopathic membranous nephropathy (iMN)

DETAILED DESCRIPTION:
To date, the first-line immunosuppressive immunosuppressive therapy of iMN includes corticosteroids combined with cyclophosphamide or rituximab (RTX). In recent randomized trials (MENTOR, GEMRITUX), the long-term remission rate of RTX is about 60%, which is similar to the remission rate of cyclophosphamide combined with corticosteroids in early studies. But there is only one published randomized trial (STARMEN) comparing the efficacy of the two protocols head-to-head. In STRAMEN trial, the long-term remission rate of cyclophosphamide+corticosteroids group was 83%, which was significantly higher than the that (58%) of the tacrolimus-RTX group. But in STRAMEN trial, only one single dose of RTX was given which might influence the efficacy of the tacrolimus-RTX arm. Therefore, head-to-head comparison of RTX (more than one dose) and cyclophosphamide+corticosteroid is needed. The optimal dose of RTX in the treatment of iMN is unclear. In MENTOR trial, RTX was given 1g on D1 and D15, and the rate of complete remission at 6 month was 0, so RTX was repeated at 6 month. Based on the experience of our center, most patients need at least one repeated dose of RTX at 6 month.

Based on the previous rationale, the investigators designed this study to compare the efficacy of cyclophosphamide plus corticosteroids with RTX in the treatment of iMN.

ELIGIBILITY:
Inclusion Criteria:

* idiopathic membranous nephropathy
* Female, must be post-menopausal, sterile or have effective contraception
* must be off steroid or mycophenolate mofetil for >1 month and alkylating agents for or RTX> 6 months
* Angiotensin-converting-enzyme inhibitor (ACEI) or angiotensin receptor blocker (ARB) for ≥ 3 months with controlled blood pressure prior to beginning of immunosuppressive therapy or if patients are intolerant to ACEI/ARB.
* proteinuria ≥4g/24h and decreased ≤ 50% from baseline

Exclusion Criteria:

* presence of active infection or a secondary cause of membranous nephropathy
* proteinuria associated with diabetic nephropathy
* pregnancy or breast feeding
* history of resistance to rituximab or alkylating agents or corticosteroid
* Patients who previously achieved remission after treatment of rituximab or alkylating agents but relapsed off rituximab or alkylating agents after 6 months are eligible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
complete or partial remission on 24 month | 24 months
  Complete remission is defined as urine protein < 0.5g/24h and serum albumin≥ 3.5g/dl. Partial remission is defined as reduction in urine protein≥50% plus urine protein ≤3.5g/24h but >0.5g/24h

SECONDARY OUTCOMES:
complete or partial remission on 6, 12 and 18 month | 6, 12 and 18 months
  complete or partial remission on 6, 12 and 18 month
complete remission on 6, 12, 18 and 24 month | 6, 12, 18 and 24 months
  complete remission on 6, 12, 18 and 24 month
time to complete or partial remission | from date of treatment until the date of first documented remission, up to 24 months
  time to complete or partial remission
change of estimated glomerular filtration rate (eGFR) | 24 months
  change of estimated glomerular filtration rate (eGFR) from baseline
serum creatinine increase ≥50 percent from baseline | 24 months
  proportion of patients with increase of serum creatinine ≥50 percent from baseline
rate of relapse | 12, 18, 24 months
  proportion of patients with relapse. Relapse is defined as development of urine protein >3.5g/24h following complete or partial remission.
anti-PLA2R levels | baseline and 3, 6, 9, 12, 18, 24 months
  Auto-antibody to the M-type phospholipase A2 receptor (PLA2R)
CD19+ B cell count | baseline and 3, 6, 9, 12, 18, 24 months
  CD19+ B cell count
Adverse events | through the study completion until 24 months
  Adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qin, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Polanco N, Gutierrez E, Covarsi A, Ariza F, Carreno A, Vigil A, Baltar J, Fernandez-Fresnedo G, Martin C, Pons S, Lorenzo D, Bernis C, Arrizabalaga P, Fernandez-Juarez G, Barrio V, Sierra M, Castellanos I, Espinosa M, Rivera F, Oliet A, Fernandez-Vega F, Praga M; Grupo de Estudio de las Enfermedades Glomerulares de la Sociedad Espanola de Nefrologia. Spontaneous remission of nephrotic syndrome in idiopathic membranous nephropathy. J Am Soc Nephrol. 2010 Apr;21(4):697-704. doi: 10.1681/ASN.2009080861. Epub 2010 Jan 28. PMID 20110379
- [Background] Dahan K, Debiec H, Plaisier E, Cachanado M, Rousseau A, Wakselman L, Michel PA, Mihout F, Dussol B, Matignon M, Mousson C, Simon T, Ronco P; GEMRITUX Study Group. Rituximab for Severe Membranous Nephropathy: A 6-Month Trial with Extended Follow-Up. J Am Soc Nephrol. 2017 Jan;28(1):348-358. doi: 10.1681/ASN.2016040449. Epub 2016 Jun 27. PMID 27352623
- [Background] Fervenza FC, Appel GB, Barbour SJ, Rovin BH, Lafayette RA, Aslam N, Jefferson JA, Gipson PE, Rizk DV, Sedor JR, Simon JF, McCarthy ET, Brenchley P, Sethi S, Avila-Casado C, Beanlands H, Lieske JC, Philibert D, Li T, Thomas LF, Green DF, Juncos LA, Beara-Lasic L, Blumenthal SS, Sussman AN, Erickson SB, Hladunewich M, Canetta PA, Hebert LA, Leung N, Radhakrishnan J, Reich HN, Parikh SV, Gipson DS, Lee DK, da Costa BR, Juni P, Cattran DC; MENTOR Investigators. Rituximab or Cyclosporine in the Treatment of Membranous Nephropathy. N Engl J Med. 2019 Jul 4;381(1):36-46. doi: 10.1056/NEJMoa1814427. PMID 31269364
- [Background] van den Brand JAJG, Ruggenenti P, Chianca A, Hofstra JM, Perna A, Ruggiero B, Wetzels JFM, Remuzzi G. Safety of Rituximab Compared with Steroids and Cyclophosphamide for Idiopathic Membranous Nephropathy. J Am Soc Nephrol. 2017 Sep;28(9):2729-2737. doi: 10.1681/ASN.2016091022. Epub 2017 May 9. PMID 28487395
- [Background] Fernandez-Juarez G, Rojas-Rivera J, Logt AV, Justino J, Sevillano A, Caravaca-Fontan F, Avila A, Rabasco C, Cabello V, Varela A, Diez M, Martin-Reyes G, Diezhandino MG, Quintana LF, Agraz I, Gomez-Martino JR, Cao M, Rodriguez-Moreno A, Rivas B, Galeano C, Bonet J, Romera A, Shabaka A, Plaisier E, Espinosa M, Egido J, Segarra A, Lambeau G, Ronco P, Wetzels J, Praga M; STARMEN Investigators. The STARMEN trial indicates that alternating treatment with corticosteroids and cyclophosphamide is superior to sequential treatment with tacrolimus and rituximab in primary membranous nephropathy. Kidney Int. 2021 Apr;99(4):986-998. doi: 10.1016/j.kint.2020.10.014. Epub 2020 Nov 7. PMID 33166580
- [Background] Dahan K, Johannet C, Esteve E, Plaisier E, Debiec H, Ronco P. Retreatment with rituximab for membranous nephropathy with persistently elevated titers of anti-phospholipase A2 receptor antibody. Kidney Int. 2019 Jan;95(1):233-234. doi: 10.1016/j.kint.2018.08.045. No abstract available. PMID 30606419